CLINICAL TRIAL: NCT01606670
Title: A Multicenter, Non-interventional Study With Neupro® to Evaluate the Perception of Pain Associated With Idiopathic Parkinson's Disease
Brief Title: Observational Study With Neupro® to Evaluate the Patient´s Perception of Pain Associated With Parkinson´s Disease
Acronym: NEUPAD
Status: Completed | Type: Observational
Sponsor: UCB Pharma GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: SP1058
Record Dates: First submitted 2012-05-22; First posted 2012-05-28 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro®
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neupro® Treatment: Routine treatment with Neupro® (2, 4, 6, 8, 10, 12, 14, 16 mg/24 h) as per approved label in the EU, which is applicable in the EU member state Germany.

SUMMARY:
The primary objective of this study is to evaluate the perception of pain associated with Parkinson´s Disease in patients who receive Neupro® for the first time.

ELIGIBILITY:
Inclusion Criteria:

* The decision by the treating physician to treat a patient with Neupro® for the first time is made before the patient's participation in this Non-Interventional Study (NIS)
* A Patient Data Consent form is signed and dated by the patient
* Male and female patients that suffer from pain associated with idiopathic Parkinson's Disease according to the physician's assessment
* Patients have not been treated with Rotigotine in the past

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pain associated with idiopathic Parkinson´s Disease. Every consecutive, eligible patient to be treated with Neupro® as per physician's decision.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (27):
- Austria (2):
  - 61, Feldbach
  - 60, Linz
- Germany (25):
  - 16, Altenholz
  - 5, Alzenau in Unterfranken
  - 22, Bad Honnef
  - 26, Bad Krozingen
  - 10, Berlin
  - 20, Cologne
  - 4, Dresden
  - 34, Düsseldorf
  - 38, Erbach im Odenwald
  - 24, Freiburg im Breisgau
  - 1, Gera
  - 3, Göttingen
  - 32, Hamburg
  - 2, Heidenheim
  - 11, Königsbrück
  - 15, Mühldorf
  - 33, Münster
  - 35, Osnabrück
  - 31, Rüsselsheim am Main
  - 7, Schriesheim
  - 44, Senftenberg
  - 12, Stadtroda
  - 13, Ulm
  - 41, Westerstede
  - 37, Würzburg

REFERENCES:
- [Result] Timmermann L, Oehlwein C, Ransmayr G, Frohlich H, Will E, Schroeder H, Lauterbach T, Bauer L, Kassubek J. Patients' perception of Parkinson's disease-associated pain following initiation of rotigotine: a multicenter non-interventional study. Postgrad Med. 2017 Jan;129(1):46-54. doi: 10.1080/00325481.2017.1258953. Epub 2016 Nov 24. PMID 27883297
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll subjects in May 2012. Overall, 28 sites enrolled 93 patients in this study.
Pre-assignment Details: Participant Flow refers to the Enrolled Set (ES).
Groups:
- Neupro® Treatment: Routine treatment with Neupro® (2, 4, 6, 8, 10, 12, 14, 16 mg/24 h) as per approved label in the EU, which is applicable in the EU member states Germany and Austria.
Period: Overall Study
Arm/Group | Neupro® Treatment
Started | 93
Safety Set | 93
Full Analysis Set | 70
Completed | 77
Not Completed | 16
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Other Reason | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set, including all enrolled patients who had applied the rotigotine transdermal patch at least once.
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 48
Region of Enrollment [Number; unit: participants]
  Austria | 6
  Germany | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit 2 in the Sum Score Calculated From the 4 Items of the Affective Dimension of the Pain Description List (Schmerzbeschreibungsliste SBL, Question 10) of the German Pain Questionnaire
Description: The Pain Description List (SBL, question 10) is part of the validated German Pain Questionnaire (DSF).
  The SBL consists of a 12 item list of adjectives. Each adjective is ranked from 0 (not applicable) to 3 (exactly applicable).
  8 of the 12 adjectives will be used to assess the sensory items of pain and 4 adjectives to describe the affective items of pain.
  The 8 sensory items are used to assess qualitative description of pain. For the 4 affective pain items, a sum score ranges from 0 (not applicable) to 12 (exactly applicable). Values above 8 can be considered noticeable.
Time Frame: From Baseline (Day 0) to Visit 2 (after at least 4 weeks on a maintenance dose of Neupro®)
Population: Full Analysis Set (FAS). The FAS includes all enrolled patients who had applied the rotigotine transdermal patch at least once and for whom valid data for the primary effectiveness variable were available from Baseline and a subsequent routine visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 70
units on a scale | -1.3 (2.8)

2. Secondary Outcome: Change From Baseline to Visit 2 in the Sum Score of the Unified Parkinson's Disease Rating Scale (UPDRS) Part II
Description: The UPDRS is a scale for the assessment of function in Parkinson's disease. Part II measures 'Activities of Daily Living'. It consists of 13 questions, each ranging from 0 (none) to 4 (severe abnormalities). The sum score of the UPDRS Part II ranges from 0 (normal) to 52 (worst score possible).
Time Frame: From Baseline (Day 0) to Visit 2 (after at least 4 weeks on a maintenance dose of Neupro®)
Population: Of the 70 patients in the Full Analysis Set (FAS), 68 patients had complete data for UPDRS Part II and are included in the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 68
units on a scale | -1.3 (4.3)

3. Secondary Outcome: Change From Baseline to Visit 2 in the Sum Score of the Unified Parkinson's Disease Rating Scale (UPDRS) Part III
Description: The UPDRS is a scale for the assessment of function in Parkinson's disease. Part III measures 'Motor Function'. It consists of 14 items with 27 questions, each ranging from 0 (normal) to 4 (severe abnormalities). The sum score of the UPDRS Part III ranges from 0 (normal) to 108 (worst score possible).
Time Frame: From Baseline (Day 0) to Visit 2 (after at least 4 weeks on a maintenance dose of Neupro®)
Population: Of the 70 patients in the Full Analysis Set (FAS), 67 patients had complete data for UPDRS Part III and are included in the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 67
units on a scale | -3.9 (7.6)

4. Secondary Outcome: Change From Baseline to Visit 2 in the Sum Score of the Unified Parkinson's Disease Rating Scale (UPDRS) Parts II+III
Description: The UPDRS is a scale for the assessment of function in Parkinson's disease. Part II measures 'Activities of Daily Living' and Part III 'Motor Function'. They consist of 40 questions, each ranging from 0 (normal) to 4 (severe abnormalities). The sum score of the UPDRS Part II+III ranges from 0 (normal) to 160 (worst score possible).
Time Frame: From Baseline (Day 0) to Visit 2 (after at least 4 weeks on a maintenance dose of Neupro®)
Population: Of the 70 patients in the Full Analysis Set (FAS), 68 patients had complete data for UPDRS Part II and 67 patients had complete data for UPDRS Part III. Thus, of the 70 patients in the FAS, 67 patients are included in the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 67
units on a scale | -5.3 (10.5)

5. Secondary Outcome: Change From Baseline to Visit 2 in the Short-form Parkinson's Disease Questionnaire (PDQ-8) Total Score
Description: The PDQ-8 is a self-administered 8 item questionnaire that assesses the overall health status. The questions will be rated from 0 (never) to 4 (always [or cannot do at all]). The total score ranges from 0 (never) to 32 (always [or cannot do at all]) with lower scores indicating a better health status.
Time Frame: From Baseline (Day 0) to Visit 2 (after at least 4 weeks on a maintenance dose of Neupro®)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 70
units on a scale | -2.0 (4.8)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the whole study from Visit 1 (Day 0) to Visit 2 (after at least 4 weeks on a maintenance dose of Neupro).
Description: Since this was a NIS with no safety objectives, only the related adverse events (AEs), ie, adverse drug reactions (ADRs), were documented.
Arm/Group | Neupro® Treatment
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 10/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neupro® Treatment (N=93)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
APPLICATION SITE ERYTHEMA (General disorders) | 1 (1)
APPLICATION SITE HYPERSENSITIVITY (General disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
GENERALISED ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days